CLINICAL TRIAL: NCT06890988
Title: Effectiveness of Comprehensive Ending the Epidemic (ETE) Interventions in the Dental Setting
Brief Title: Ending the Epidemic Interventions in the Dental Setting - UH3
Acronym: ETE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Michael Yin, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAT8854 - UH3; 4UH3DE031258 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-03-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection
Keywords: clinical decision support; acceptability; feasibility; implementation science; HIV testing

STUDY DESIGN:
Intervention Model Description: Sites will be randomized to one of 2 arms: (AB) Standard Dental Care Team model followed by crossover to an Enhanced Dental Care Team model with a Care Navigator, or (BA) Enhanced Dental Care Team model with a Care Navigator followed by crossover to a Standard Dental Care Team model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Dental Care Team model (Placebo Comparator): Multicomponent HIV Service Package delivered without a Care Navigator
  Interventions: Other: Multicomponent HIV Service Package
- Enhanced Dental Care Team model with a Care Navigator (Experimental): Multicomponent HIV Service Package delivered with a Care Navigator
  Interventions: Other: Care Navigator; Other: Multicomponent HIV Service Package

INTERVENTIONS:
Other: Care Navigator — The Care Navigator will be added to the dental team as an added resource to:
  1. Champion the use of the multicomponent HIV intervention in the dental clinic among clinic administrators, residents, dental hygienists, dental assistants, and other dental team staff.
  2. Provide technical assistance
  3. Provide logistical assistance ; and
  4. Support dental team in educating patients about HIV prevention and treatment options
  Arms: Enhanced Dental Care Team model with a Care Navigator
Other: Multicomponent HIV Service Package — Multicomponent HIV Service Package consisting of:
  1. Clinical Decision Support (CDS) within electronic medical record (EMR) system to help providers identify patients who would benefit from HIV screening or re-engagement in HIV care.
  2. Point-of-care HIV testing in the dental clinic.
  3. Patient and provider-facing educational materials to support providers in discussing HIV prevention options (for patients who test HIV negative) and treatment (for patients who test HIV positive or are out of HIV care) options.

SUMMARY:
The purpose of this study is to use information technology (IT) to support the efficient delivery of HIV prevention and care best practices in the dental care setting.

DETAILED DESCRIPTION:
Routine preventative HIV screening in all health care settings is considered a best practice by the Centers for Disease Control and Prevention (CDC), Department of Health and Human Services (DHHS) Ending the Epidemic (ETE) Initiative, the New York State Blueprint to End the AIDS Epidemic. Despite this, many patients are not screened for HIV during routine care, including in dental care settings, resulting in missed opportunities for identifying undiagnosed HIV infections and providing education for pre-exposure prophylaxis (PrEP). This study will use information technology to support the delivery of HIV prevention and care best practices in the dental care setting. Dental residents will receive a Best Practice (BPA) alert whenever they have a patient who should be offered HIV screening. This BPA is linked to an order set to simplify ordering HIV tests and reporting results.

A critical knowledge gap for implementing these ETE activities in the dental setting is whether comprehensive ETE efforts could be integrated into existing dental teams consisting of practitioners, dental assistants and hygienists or require augmentation by a dedicated care navigator. To evaluate these two models, the investigators will conduct a crossover clinical trial in 3 urban general dentistry programs (NYP-Columbia, NYP-Cornell, NYP-Queens) randomized to one of 2 arms: (AB) Standard Dental Care Team model followed by crossover to an Enhanced Dental Care Team model with a Care Navigator, or (BA) Enhanced Dental Care Team model with a Care Navigator followed by crossover to a Standard Dental Care Team model.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Dental Team (Provider, Hygienist, Dental Assistant, Care Navigator) at one of the randomized sites with direct patient contact
* Able to provide written informed consent.

Exclusion Criteria:

- Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that complete point of care HIV testing out of patient encounters receiving clinical decision support (CDS) prompts for HIV testing | 10 months after start of each arm
  Proportion of patients receiving clinical decision support (CDS) prompts for HIV testing that complete point of care HIV testing over the intervention period under the Enhanced versus Standard Dental Care Models.

SECONDARY OUTCOMES:
Provider acceptability of multicomponent HIV service package in dental clinics | 5-10 months after start of each arm
  Provider acceptability of multicomponent HIV service package in dental clinics under the Enhanced versus Standard Dental Care Models. Acceptability will be assessed using the validated Acceptability of Intervention Measure (AIM). AIM is a 4-item scale where respondents rate each item using a 5-point ordinal scale that ranges from "completely disagree=1" to "completely agree=5". The AIM is scored by averaging responses across the 4 items. A higher average score indicates greater acceptability, which is a better outcome.
Provider feasibility of multicomponent HIV service package in dental clinics | 5-10 months after start of each arm
  Provider feasibility of multicomponent HIV service package in dental clinics under the Enhanced versus Standard Dental Care Models. Feasibility will be assessed using the validated Feasibility of Intervention Measure (FIM). FIM is a 4-item scale where respondents rate each item using a 5-point ordinal scale that ranges from "completely disagree=1" to "completely agree=5". The FIM is scored by averaging responses across the 4 items. A higher average score indicates greater acceptability, which is a better outcome.
Proportion of patients receiving CDS prompt for HIV testing that complete subsequent HIV testing outside of the dental clinic | Within 12 months following dental visit
  Proportion of patients receiving CDS prompt for HIV testing that complete subsequent HIV testing outside of the dental clinic under the Enhanced versus Standard Dental Care Models.
Proportion of patients receiving CDS prompt for HIV testing with subsequent appointment at an HIV prevention clinic | Within 12 months following dental visit
  Proportion of patients receiving CDS prompt for HIV testing with subsequent appointment at an HIV prevention clinic under the Enhanced versus Standard Dental Care Models.
Proportion of patients receiving CDS prompt for HIV testing subsequently prescribed pre-exposure prophylaxis (PrEP) medication | Within 12 months following dental visit
  Proportion of patients receiving CDS prompt for HIV testing subsequently prescribed pre-exposure prophylaxis (PrEP) medication under the Enhanced versus Standard Dental Care Models.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York
  - Weill Cornell Medical Center / NewYork-Presbyterian Hospital, New York, New York
  - NYP-Queens, Queens, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be shared with other researchers within Columbia University at the discretion of the Principal Investigator, and only when the Institutional Review Board (IRB) approval has been granted to allow for the sharing of such data.